CLINICAL TRIAL: NCT05565690
Title: Diagnostic Yield of Preoperative Magnetic Resonance Spectroscopy for Solitary Intra-axial Brain Lesion in Comparison to Histopathology
Brief Title: Role of MRS in Brain Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Aboelmagd Ahmed, Resident doctor, Assiut University
Other Study IDs: MRS in brain lesions
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Brain Lesion (General); Mrs
MeSH Terms: conditions — Melkersson-Rosenthal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRS — It is a tool used to determine the molecular structure of compounds or to detect the compound presence , it provides metabolic information from living brain

SUMMARY:
Aim of the study is evaluation of accuracy of magnetic resonance spectroscopy in differentiation between neoplastic and non neoplastic lesions and determination the type of neoplasm

DETAILED DESCRIPTION:
The annual global age-standardized incidence of primary malignant brain tumors is ~3.7 per 100,000 for males and 2.6 per 100,000 for females . Rates appear to be higher more in developed countries (males, 5.8 and females, 4.1 per 100,000) than in less developed countries (males 3.0 and females 2.1 per 100,000). More than half of all brain tumors are Intraparenchymal . Diagnosis of brain lesions and other focal intracranial lesions based on imaging methods alone is still facing a challenging problem. Accurate diagnosis is fundamentally vital for clinical management in patients with brain tumors. CT and standard MRI are the first line imaging modalities in evaluation of brain lesions; however, it does not always provide more precise details and characterization of the lesions whether it is benign or malignant. Conventional imaging techniques do not provide exact information about vascularity, cellularity and metabolism of the mass lesion . Magnetic Resonance Spectroscopy (MR Spectroscopy) is one of the tools used to determine themolecular structures of compounds or to detect the compound presence. MR Spectroscopy provides metabolic information from living tissues. The major brain metabolites detected are choline, creatine, N-acetyl aspartate (NAA), lactate, myoinositol, glutamine, glutamate, lipids and the amino acids leucine and alanine. Brain lesions show abnormal values of these metabolites as compared to normal tissue.Our study aims to determine the accuracy of MRS in differentiation between neoplastic and non neoplastic lesions and determination the type of neoplasm, Discriminating neoplastic from non-neoplastic brain lesions is extremely necessary since a misdiagnosis can lead to a severe effect on neurosurgery and exposure to toxic chemotherapy or radiotherapy, which may cause damage to brain tissues.

ELIGIBILITY:
Inclusion Criteria:

* patients with solitary intraaxial brain lesions
* patients with de novo lesions
* Patient age : any age

Exclusion Criteria:

* patients with multiple intra-axial brain lesions
* patients with extra-axial brain lesions
* patients with recurrent lesions
* patients receiving chemotherapy or radiotherapy
* patients unfit for surgery

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with brain lesions of any age
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of accuracy of magnetic resonance spectroscopy in differentiation between neoplastic and non neoplastic lesions and determination the type of neoplasm | Baseline
  Analysis of the MRS metabolites peaks and test if they can differentiate between neoplastic and non neoplastic lesions and grades of neoplasm by comparison with postoperative histopathology

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ahmed Abd-Elaleem, Lecturer, Study Director — Assiut University